CLINICAL TRIAL: NCT01002482
Title: Impact of the Use of a Computerized Protocol for Glucose Control Named CGAOtm on the Outcome of Critically Ill Patients
Brief Title: Computerized Glucose Control in Critically Ill Patients
Acronym: CGAO-REA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier of Chartres (Other)
Collaborators: Société Française d'Anesthésie et de Réanimation (Other); Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr Pierre KALFON, principal investigator, Centre Hospitalier of Chartres
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CGAO-REA-01
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Hyperglycemia; Critical Illness
Keywords: Hyperglycemia; Hypoglycemia; Intensive Care Unit; Glucose Control; Insulin; Computer Protocol; Metabolic Disorders
MeSH Terms: conditions — Hyperglycemia; Critical Illness; Hypoglycemia; Insulin Resistance; Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CGAO-based Glucose Control (Experimental): Use of a Computerized Protocol fot Tight Glycemic Control named CGAO software in order to maintain Blood Glucose Levels between 4.4 and 6.1 mmol/l.
  Interventions: Device: CGAO-based Glucose Control
- Standard-Care Glucose Gontrol (Active Comparator): Use of Standard-Care Methods for Glucose Control targeting Blood Glucose Levels inferior to 10 mmol/l.
  Interventions: Device: Standard-Care Glucose Control

INTERVENTIONS:
Device: CGAO-based Glucose Control — Use of a clinical computerized decision-support system named CGAOtm designed to achieve tight glucose control in various ICU settings, and fine-tuned to reduce glucose variability without increasing the incidence of severe hypoglycemia or nurse workload.
  CGAOtm is based on explicit replicable recommendations following each blood glucose measurement for insulin rates and time to next measurement, and reminders, alerts, graphic tools, trends, and individual on-line data aimed at increasing confidence of the nursing staff in the computer protocol and giving care staff a method for controlling the process during the whole ICU stay, according to a "human-in-the-loop" approach.
  The algorithm used in the CGAOtm software for the calculation of the recommended insulin rates derived from a PID (Proportional-integral-derivative) controller, a generic control loop feedback mechanism widely used in industrial control.
  Other Names: CGAO, LC_CGAO version1
  Arms: CGAO-based Glucose Control
Device: Standard-Care Glucose Control — Patients in the control group will receive conventional insulin therapy using the "usual care" protocol of each participating centre (already used in the centre before the beginning of the trial and targeting blood glucose levels inferior to 180 mg/dl).
  Other Names: Usual care
  Arms: Standard-Care Glucose Gontrol

SUMMARY:
The aim of the study is to determine whether the use of the CGAOtm software is associated with a decrease in 90-day mortality when compared with the use of standard care methods for glucose control with target blood glucose levels inferior to 180 mg/dl. The CGAOtm software is designed to assist physicians and nurses in achieving tight glucose control (defined by a target for blood glucose levels between 80 and 110 mg/dl) in critically ill patients.

DETAILED DESCRIPTION:
Hyperglycemia in response to critical illness has long been associated with adverse outcomes.

In 2001, the first "Leuven study", a randomized controlled trial conducted in surgical intensive care patients comparing a strategy based on a nurse-driven protocol for insulin therapy in order to maintain normal blood glucose levels [80 - 110 mg/dl] with standard care defined at the time as intravenous insulin started only when blood glucose level exceeded 215 mg/dl and then adjusted to keep blood glucose level between 180 and 200 mg/dl, showed a reduction in hospital mortality by one third.

The results of this trial have been enthusiastically received and rapidly incorporated into guidelines, such as the Surviving Sepsis Campaign in 2004, and now endorsed internationally by numerous professional societies.

However, subsequent randomized controlled trials have failed to confirm a mortality benefit with intensive insulin therapy among critically ill patients, in whom stress hypoglycemia is common. Moreover the Normoglycemia in Intensive Care Evaluation - Survival Using Glucose Algorithm Regulation (NICE-SUGAR) study, an international multicentre trial involving 6104 patients, the largest trial of insulin therapy to date, showed a lower 90-day mortality in the control group targeted blood glucose levels inferior to 180 mg/dl when compared to the intervention group with tight glucose control [80 - 110 mg/dl].

In addition, many studies and meta-analyses have reported high rates of hypoglycemia with tight glucose control. Consequently, considerable controversy has emerged as to whether tight glucose control is warranted in all critically ill patients especially as tight glucose control (without appropriate computer protocol) causes a significant increase in nurse workload.

The conflicting results between the first Leuven study and the NICE-SUGAR study could be explained by numerous differences between the two trials : the specific method (algorithms, compliance of nurses and physicians with recommendations, etc) used to achieve tight glucose control in each randomized control trial could be a major issue.

Several experimental and observational studies have highlighted the possible negative impact of glucose variability (large fluctuations in blood glucose possibly with undetected hypoglycemia and hypokalemia alternating with hyperglycemia) when implementing tight glucose control, be it due to the intrinsic properties of the algorithms used, technical factors (errors in measurements of the blood glucose level or lack of control over intravenous insulin therapy) or human factors (delay in performing glucose measurements or non respect of recommendations not based on clinical expertise but as a consequence of insufficient training inducing a lack of confidence in the algorithms by inexperienced nurses).

Therefore, remaining concerns about the best way to achieve glucose control in the ICU reduce the impact of conclusions of all of the recent randomized controlled trials on tight glucose control : are the negative results due to the concept, tight glucose control with intensive insulin therapy in critically ill patients in order to reduce the toxicity of high blood glucose levels, or are the negative results mainly due to specific methods used for achieving tight glucose control ? In most cases the methods used in clinical trials were never tested in numerical patients according to existing and validated models (in SILICO expertise) before implementing them in clinical practice on real patients.

Particularly, whether the use of a clinical computerized decision-support system (CDSS) designed for achieving tight glucose control in various ICU settings, and fine-tuned to reduce glucose variability, without increasing the incidence of severe hypoglycemia nor the nurse workload, has an impact on the outcome of patients staying at least three days in an ICU remains to be tested.

Among the different CDSS, the CGAOtm software has been developed to standardize different aspects of glucose control in an ICU setting based on 1) explicit replicable recommendations following each blood glucose level measurement concerning insulin rates and time to next measurement, 2) reminders and alerts and 3) various graphic tools, trends, and individual on-line data aiming to increase the confidence of the nursing staff in the computer protocol and therefore their adherence, to reduce necessary training time, and to give physicians and nurses a way to control the tight glucose control process during the whole ICU stay. Moreover, the CGAOtm software is designed to take into account irregular sampling, saturations, and some precision and stability issues.

The aim of the study is to evaluate the capability of the CGAOtm software to reduce 90-day mortality in a mixed ICU population of patients requiring intensive care for at least three days.

Sample size and power calculations. The expected all cause 90-day mortality in the control group is 25 % (identical to the observed all cause 90-day mortality in the control group of the NICE-SUGAR trial). Considering that all cause 90-day mortality in the experimental group (computer protocol group) is expected to be 22 % (absolute reduction of 3 %), considering an alpha risk and a beta risk respectively of 0.05 and 0.20 and three intermediate analyses performed according to the O'Brien-Fleming design, 3,211 patients per treatment arms are needed and will be recruited from the participating 60 centres, all located in France.

ELIGIBILITY:
Inclusion Criteria:

* At time of the patient's admission to the ICU, the treating ICU specialist expects the patient will require treatment in the ICU that extends beyond the calendar day following the day of admission.

Exclusion Criteria:

* Age < 18 years or patient under guardianship.
* Pregnancy.
* Moribund patient or imminent death in the ICU (e.g. patient expected to die in the ICU within 24 hours).
* At time of the patient's admission, the treating physicians are not committed tu full supportive care.
* Patient admitted to the ICU for treatment of diabetic ketoacidosis or hyperosmolar state.
* Patient admitted to the ICU for hypoglycemia.
* Patient thought to be at abnormally high risk of suffering hypoglycemia (e.g. known insulin secreting tumor or history of unexplained or recurrent hypoglycemia or fulminant hepatic failure).
* Patient who have suffered hypoglycemia without documented full neurological recovery
* Patient is expected to be eating before the end of the day following admission.
* Patient previously enrolled in the CGAO-REA study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2684 (Actual)
Dates: Start 2009-10; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Kalfon, MD, Principal Investigator — Centre Hospitalier de Chartres; Bruno Riou, MD PhD, Study Director — G.H.U. Est, C.H.U. Pitié-Salpétriêre; Djillali Annane, MD PhD, Study Chair — G.H.U. Ouest, Hôpital Raymond Poincaré; Jean Chastre, MD PhD, Study Chair — G.H.U. Est, Pitié-Salpétriêre; Pierre-François Dequin, MD PhD, Study Chair — CHRU TOURS; Hervé Dupont, MD PhD, Study Chair — CHRU Amiens; Carole Ichai, MD PhD, Study Chair — CHRU de Nice; Yannick Malledant, MD PhD, Study Chair — CHRU Rennes; Philippe Montravers, MD PhD, Study Chair — G.H.U. Nord Bichat-Claude Bernard
Locations (35):
- France (35):
  - C.H.U. Hôpital Nord, Amiens
  - C.H. d'Avignon, Avignon
  - G.H.U. Nord Hôpital Jean Verdier, Bondy
  - Polyclinique Jean Vilar, Bruges
  - Hôpital Sainte-Camille, Bry-sur-Marne
  - C.H. de Chartres, Chartres
  - C.H. Châteauroux, Châteauroux
  - Hôpital Sud-Francilien - Site Corbeil, Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - C.H. Victor Jousselin, Dreux
  - Raymond Poincaré, Garches
  - Centre Hospitalier Départemental Les Oudairies, La Roche-sur-Yon
  - G.H.U. Sud Bicêtre, Le Kremlin-Bicêtre
  - Hôpital de Mantes-La-Jolie, Mantes-la-Jolie
  - Hôpital Paul Desbief, Marseille
  - C.H.U. La Timone, Marseille
  - Hôpital Ambroise Paré, Marseille
  - C.H.U. de -Hôpital Saint-Eloi, Montpellier
  - C.H.U. Lapeyronie, Montpellier
  - C.H.U. Nantes - Hôpital Laennec, Nantes
  - C.H.U. de Nice - Hôpital Saint-Roch, Nice
  - Hôpital Européen Georges Pompidou, Paris
  - G.H.U. Pitié-Salpétriêre, Paris
  - Institut Mutualiste Montsouris, Paris
  - G.H.U. Nord Claude Bernard, Paris
  - C.H. de Pau, Pau
  - CHU de Bordeaux - Groupe Hospitalier Sud, Hôpital Haut Lévêque, Pessac
  - C.H. René Dubos, Pontoise
  - C.H. Bourran, Rodez
  - C.H.U. Hôpitaux de Rouen, Rouen
  - Hôpital Foch, Suresnes
  - C.H. Intercommunal - Hôpital Font-Pré, Toulon
  - C.H.U. Purpan, Toulouse
  - C.H.U. Rangueil, Toulouse
  - C.H.R.U. de Tours, Tours

REFERENCES:
- [Background] Carli P, Martin C. [Impact of Nice-Sugar: is there a need for another study on intensive glucose control in ICU?]. Ann Fr Anesth Reanim. 2009 Jun;28(6):519-21. doi: 10.1016/j.annfar.2009.05.002. Epub 2009 Jun 4. No abstract available. French. PMID 19500942
- [Background] Guerrini A; Roudillon G; Gontier O; Rebaï L; Isorni MA; Mutinelli-Szymanski P; Sorine M; Kalfon P. High glycemic variability induced by inappropriate algorithms for intensive insulinotherapy: the example of the NICE-SUGAR study. Abstract award winners: The best pre-selected abstracts of the 22th Annual Congress of the European Society of Intensive Care Medicine, 11-14 October 2009, Vienna, Austria. Intensive Care Med. 2009 Sep;35 Suppl 1:S111.
- [Background] Gontier O; Hamrouni M; Lherm T; Monchamps G; Ouchenir A; Kalfon P. The CGAO software improves glycaemic control in intensive care patients without increasing the incidence of severe hypoglycaemia nor the nurse workload. Abstracts of the 21th Annual Congress of the European Society of Intensive Care Medicine, 21-24 September 2007, Lisbon, Portugal. Intensive Care Med. 2008 Sep;34 Suppl 2:S220.
- [Background] Abstracts of the 20th Annual Congress of the European Society of Intensive Care Medicine, 7-10 October 2007, Berlin, Germany. Intensive Care Med. 2007 Sep;33 Suppl 2:S5-271. No abstract available. PMID 18183643
- [Derived] Kalfon P, Le Manach Y, Ichai C, Brechot N, Cinotti R, Dequin PF, Riu-Poulenc B, Montravers P, Annane D, Dupont H, Sorine M, Riou B; CGAO-REA Study Group. Severe and multiple hypoglycemic episodes are associated with increased risk of death in ICU patients. Crit Care. 2015 Apr 8;19(1):153. doi: 10.1186/s13054-015-0851-7. PMID 25888011
- [Derived] Kalfon P, Giraudeau B, Ichai C, Guerrini A, Brechot N, Cinotti R, Dequin PF, Riu-Poulenc B, Montravers P, Annane D, Dupont H, Sorine M, Riou B; CGAO-REA Study Group. Tight computerized versus conventional glucose control in the ICU: a randomized controlled trial. Intensive Care Med. 2014 Feb;40(2):171-181. doi: 10.1007/s00134-013-3189-0. Epub 2014 Jan 14. PMID 24420499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients who were assumed to require at least 3 days in the ICU were eligible for inclusion. The study, carried out between October 2009 and June 2011, involved 34 ICUs (19 in academic tertiary care hospitals and 15 in community hospitals)
Pre-assignment Details: 876 participants were eligible but were excluded: 844 Had objection of the treating physician, 32 declined to participate
Period: Overall Study
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Started | 1351 | 1333
Completed | 1336 | 1312
Not Completed | 15 | 21
Not completed — Withdrawal by Subject | 14 | 21
Not completed — Included twice | 1 | 0

BASELINE CHARACTERISTICS:
Population: Among the 2684 randomized patients, 1351 were assigned to tight computerized glucose control and 1333 to conventional glucose control. Thirty six patients were discarded from any analysis, 35 because they withdrew consent and 1 because he/she was included twice. Baseline analysis was performed only for the 2648 included and not discarded patients.
Groups:
- Total: Total of all reporting groups
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol | Total
Number analyzed (Participants) | 1336 | 1312 | 2648
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 720 | 722 | 1442
  >=65 years | 616 | 590 | 1206
Age Continuous [Mean (Standard Deviation); unit: years] | 61.5 (16.2) | 61.6 (16.2) | 61.5 (16.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 474 | 468 | 942
  Male | 862 | 844 | 1706
Region of Enrollment [Number; unit: participants]
  France | 1336 | 1312 | 2648

OUTCOME MEASURES:

1. Primary Outcome: All-cause 90-day Mortality
Time Frame: Day 90
Measure: Number; unit: participants
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
participants | 431 | 447

2. Secondary Outcome: All-cause 28-day Mortality
Time Frame: Day 28
Measure: Number; unit: participants
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
participants | 326 | 328

3. Secondary Outcome: All-cause Intensive Care Unit Mortality
Time Frame: Date of discharge from the ICU
Measure: Number; unit: participants
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
participants | 302 | 310

4. Secondary Outcome: All-cause In-hospital Mortality
Time Frame: Day of discharge from the hospital
Measure: Number; unit: participants
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
participants | 376 | 393

5. Secondary Outcome: Intensive Care Unit Free Days
Description: Intensive care unit free days was 28-day-ICU-free-days i.e. was calculated by subtracting the actual ICU duration in days from 28 with patients who died at day 28 or before being assigned 0 free-days and those who had a stay in ICU of 28 days or more being also assigned 0 free-days
Time Frame: 28 days
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
days | 14 [0 to 22] | 13 [0 to 23]

6. Secondary Outcome: Time Spent in Blood Glucose Target
Time Frame: Day of discharge from the ICU
Reporting Status: Not Posted

7. Secondary Outcome: Severe Hypoglycemia
Description: Number of patients with severe biological hypoglycemia (defined as blood glucose of 40 mg per deciliter or less)regardless of clinical signs
Time Frame: Date of discharge from the ICU
Measure: Number; unit: participants
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1314 | 1289
participants | 174 | 79

8. Secondary Outcome: Hospital Length of Stay
Time Frame: Date of discharge from the hospital
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
days | 20 [10 to 37] | 20 [9 to 39]

9. Secondary Outcome: Intensive Care Unit Length of Stay
Time Frame: Date of discharge from the ICU
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Number analyzed (Participants) | 1336 | 1312
days | 9 [5 to 18] | 8 [4 to 17]

10. Secondary Outcome: Incidence of Nosocomial Bacteriemia
Time Frame: Date of discharge from the ICU
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | CGAO-based Glucose Control | Standard-Care Glucose Gontrol
Serious Adverse Events (participants affected / at risk) | 20/1336 | 6/1312
Other Adverse Events (participants affected / at risk) | 0/1336 | 0/1312
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CGAO-based Glucose Control (N=1336) | Standard-Care Glucose Gontrol (N=1312)
BG of 40 mg per deciliter or less accompanied with observed or suspected neurological symptoms (Metabolism and nutrition disorders) | 20 (23) | 6 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No